CLINICAL TRIAL: NCT01539135
Title: The Influence of Endotracheal Tube Cuff Design on Intraoperative Microaspiration and Postoperative Respiratory Complications
Brief Title: The Influence of Endotracheal Tube Design on Fluid Leakage Into the Lungs During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COVAIPR0235
Record Dates: First submitted 2012-02-06; First posted 2012-02-27 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Aspiration
Keywords: Aspiration, Respiratory
MeSH Terms: conditions — Respiratory Aspiration | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hi-Lo endotracheal tube (Active Comparator): Hi-Lo endotracheal tube with barrel shaped cuff with 20 cc of methylene blue instilled above the cuff once post intubation for the duration of the surgical procedure
  Interventions: Drug: Methylene Blue
- TaperGuard endotracheal tube (Experimental): TaperGuard endotracheal tube with taper shaped cuff with 20 cc methylene blue instilled above the cuff once post intubation for the duration of the surgical procedure
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — 20 cc methylene blue instilled above the cuff once after intubation for the duration of the surgical procedure
  Other Names: Methylene Blue Dye

SUMMARY:
Surgical patients have an endotracheal tube inserted into their windpipe to help them breathe while under general anesthesia. These tubes have a "cuff" on the outside that is inflated in the trachea to help prevent fluids from leaking into the lungs. These cuffs come in different shapes and sizes. The TaperGuard endotracheal tube has a taper-shaped cuff that has been shown in animals to decrease the leakage of fluid past the cuff better than a traditional tube that has a barrel-shaped cuff. This study is designed to examine whether the use of the TaperGuard tube during surgery on humans decreases the amount of leakage past the cuff to a greater degree than the traditional barrel-shaped cuff. In addition, the study will investigate whether the use of the TaperGuard tube is associated with a decrease in respiratory complications often seen following surgery which may be related to fluid leaking past the cuff and into the lungs. It is thought that the use of the TaperGuard endotracheal tube will result in a decrease in fluid leakage past the cuff and that it will be associated with a decrease in respiratory complications during the 30 days after surgery.

DETAILED DESCRIPTION:
This study is designed to yield data on the intraoperative use of TaperGuard™endotracheal tubes and its potential influence on postoperative pulmonary complications and outcomes. The TaperGuard Basic tube has a taper-shaped cuff and has been shown, via bench and animal testing, to decrease microaspiration, which has been associated with respiratory difficulties. The intraoperative use of this tube (i.e. during short term intubation), and its impact on postoperative complications and outcomes has not been investigated. This study will determine whether the intraoperative use of the TaperGuard tube results in a decrease in microaspiration compared to the Hi-Lo endotracheal tube having a barrel-shaped cuff. Moreover, the relationship between a decrease in microaspiration and subsequent decrease in postoperative respiratory complications will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female of all races
* Older than 18 years old
* Scheduled for an elective surgical procedure under general anesthesia for no less than 2hr and no more than 12hr with planned endotracheal intubation via the oral route
* Willing and able to give informed consent for participation in the study
* Anticipated extubation at the conclusion of general anesthesia in the operating room and prior to admission to the PACU
* Expected hospital stay of greater than or equal to 23hrs

Exclusion Criteria:

* Preexisting acute respiratory illness requiring antibiotic treatment within the two weeks prior to surgery
* Temperature of over 101 degrees F (38.3 C) at time of scheduled surgery
* Surgical requirement for naso-tracheal intubation
* Patients undergoing surgical procedures directly on the lungs, trachea, or airways
* Presence of tracheostomy
* History of allergic reaction to methylene blue
* Methemoglobinemia, glucose-6-phosphate (G6PD) deficiency
* Renal insufficiency or failure
* Requirement for prolonged intubation and/or ventilation beyond the point of PACU admission
* Intraoperative use of nitrous oxide, to avoid the increase in cuff pressure due to diffusion of gas over time
* Psychiatric drugs of the following classifications: selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), and monoamine oxidase inhibitors (MAOIs).
* Patients younger than 18 years of age
* Prone positioning during surgery
* Pregnant or lactating women based on standardized preoperative screening protocols
* Legally detained prisoner status
* Unwilling or unable to give informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Bent, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Hospital and Clinics, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Started | 43 | 37
Completed | 43 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube | Total
Number analyzed (Participants) | 43 | 37 | 80
Age, Categorical [Count of Participants; unit: Participants] — Age: >18years Gender, male, female
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 37 | 33 | 70
    >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.7) | 53.5 (14.7) | 56 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 27 | 28 | 55
Region of Enrollment [Number; unit: participants]
  United States | 43 | 37 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dye Leakage
Description: Blue dye will be instilled above the endotracheal tube cuff immediately after intubation where it will remain for the duration of the surgery. The presence of dye leakage past the endotracheal tube cuff will be determined via analysis of bronchoscopic images taken at the end of the surgical procedure when surgical closure has begun.
Time Frame: Duration of surgical procedure - from 2 to 12 hours
Measure: Number; unit: participants
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Number analyzed (Participants) | 43 | 37
participants | 3 | 2

2. Secondary Outcome: Length of Hospital Stay
Description: Time of readiness for discharge from PACU, defined as when an Aldrete score of greater than or equal to 8 is given, to the time at which discharge (from the hospital) orders are written. The inpatient period may extend up to 72 hours.
Time Frame: Time from discharge from PACU to discharge from hospital up to 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Number analyzed (Participants) | 43 | 37
hours | 42.4 (19.6) | 34.9 (16.7)

3. Secondary Outcome: Number of Participants With Postoperative Pneumonia
Description: Diagnosis of postoperative pneumonia during the 30 day follow up period after surgery
Time Frame: Up to 30 days after surgery
Measure: Number; unit: participants
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Number analyzed (Participants) | 43 | 37
participants | 1 | 0

4. Secondary Outcome: Number of Participants With Unanticipated Intensive Care Unit Admission
Description: Incidence of unscheduled Intensive Care Unit admission after surgery and length of ICU stay if applicable.
Time Frame: Time from discharge from PACU to discharge from hospital up to 72 hours
Measure: Number; unit: participants
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Number analyzed (Participants) | 43 | 37
participants | 3 | 3

ADVERSE EVENTS:
Arm/Group | Hi-Lo Endotracheal Tube | TaperGuard Endotracheal Tube
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/37
Other Adverse Events (participants affected / at risk) | 0/43 | 0/37

LIMITATIONS AND CAVEATS:
This was a feasibility study and based on the results, we do not believe that a larger, multicenter randomized controlled trial would be appropriate. The study wasn't powered to find any significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No